CLINICAL TRIAL: NCT05302726
Title: Betydning af Eksogent østrogen på Serum Kortisol Under Synacthen-stimulering Hos Hypogonade Kvinder Med Binyrebarkinsufficiens
Brief Title: Impact of Exogenous Estrogens on Cotisol Levels During Synacthen Stimulation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Mikkel Andreassen, Consultant, PhD associate professor, Rigshospitalet, Denmark
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: H-20048992
Record Dates: First submitted 2022-03-18; First posted 2022-03-31 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Adrenal Insufficiency; Hypogonadism Female
MeSH Terms: conditions — Adrenal Insufficiency | interventions — Estrogens

STUDY DESIGN:
Intervention Model Description: All patients will be examinated after 3 months on oral estrogen, 3 months on transdermal estrogen and after 3 months without estrogen substitution
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Oral estrogen (Active Comparator): oral estrogen (2 mg/24 hours)
  Interventions: Drug: Estrogen
- Transdermal estrogen (Active Comparator): Transdermal estrogen (100ug/24 hours)
  Interventions: Drug: Estrogen
- No treatment (No Intervention): Estrogen pause

INTERVENTIONS:
Drug: Estrogen — Transdermal and oral estrogen both as substitution therapy
  Arms: Oral estrogen; Transdermal estrogen

SUMMARY:
The aim is to investigate impact of exogenous estrogens on cotisol Levels during synacthen stimulation in female hypogonal patients on estrogen substitution. Both patients with and withour adrenal insufficiency will be studied

DETAILED DESCRIPTION:
The aim is to investigate impact of exogenous estrogens on cotisol levels during synacthen stimulation in female hypogonal patients on estrogen substitution. Both patients with and without adrenal insufficiency will be studied . All patients (inclusion criteria age 18-50 years, BMI <35) will be followed for 6 months and have 3 synacthentests performed: One on transdermal estrogen (minimum 3 months), one on oral estrogens (min 3 months) and one without estrogen substitution for at least 3 months. Primary endpoint is change in serum cortisol 30 minutes after synacthen stimulation

ELIGIBILITY:
Inclusion Criteria:

* Hypogonadism
* Treatment with estrogen substitution

Exclusion Criteria:

* Other formulations of glucocorticoid than oral hydrocortisone
* Pregnancy
* BMI > 35

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 20 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in serum cortisol oral estrogen | Assessment will take place before and 3 months after introduction of the intervention
  Change in serum cortisol 30 minutes after stimulation with synacthen in patients on oral estrogen vs no estrogen substitution
Change in serum cortisol transdermal estrogen | Assessment will take place before and 3 months after introduction of the intervention
  Change in serum cortisol 30 minutes after stimulation with synacthen in patients on transdermal estrogen vs no estrogen substitution

CONTACTS AND LOCATIONS:
Overall Officials: Mikkel M Andreassen, Principal Investigator — Department of endocrinology and metabolism
Locations (1):
- Mikkel Mr Andreassen, Copenhagen, Denmark